CLINICAL TRIAL: NCT05897723
Title: Safety and Efficacy of Fractional Radiofrequency for the Reduction of Surgical Scar Formation
Brief Title: Fractional Radiofrequency for Reduction of Surgical Scar Formation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI0120
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Non-randomized, single-center, split-body, evaluator blinded
Masking Description: Independent blinded evaluator assessment of the surgical scar sites using the Global Aesthetic Improvement Scale (GAIS), comparing follow-up visit photographs for for both the treated and untreated sides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): All enrolled subjects will undergo breast reduction or breast mastectomy in which scar assessment will be made after pre-surgical treatment in a split-body design, involving a single treatment of RF application to one side of the surgical area(s) within 24 hours prior to the procedure. The subject will act as their own control, where one surgical area will be treated, and the other will not be and will act as the control. Tissue samples will be biopsied from RF treated skin, as well as non-treated skin, at follow up visits. The samples will be used for histological evaluation to assess tissue structure and regeneration following surgery.
  Interventions: Device: Fractional Radiofrequency

INTERVENTIONS:
Device: Fractional Radiofrequency — Fractional Radiofrequency (RF) delivering nano-fractional RF energy, causing fractional ablation and coagulation at the treatment site.

SUMMARY:
Safety and Efficacy of Fractional Radiofrequency for the Reduction of Surgical Scar Formation

DETAILED DESCRIPTION:
The study will evaluate up to 20 subjects scheduled to undergo breast reduction or breast mastectomy in which scar assessment can be made after pre-surgical treatment in a split-body design. The study will involve a single treatment of radiofrequency (RF) applied to one side of the surgical area(s) within 24 hours prior to the procedure. The subject will act as their own control, where one surgical area will be treated, and the other will not be and will act as the control. Tissue samples will be biopsied from the RF treated skin, as well as non-treated skin, at follow up visits. The samples will be used for histological evaluation to assess tissue structure and regeneration following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female subjects 21-75 years of age who are seeking pre-treatment for the prevention of surgical scars.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Willing to avoid direct sunlight to the treatment area for the duration of the study.
5. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study, and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Subjects with any implantable metal device in the treatment area
2. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
3. Permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
4. Current or history of any kind of cancer, or dysplastic nevi.
5. Severe concurrent conditions, such as cardiac disorders.
6. Pregnancy or intending to become pregnant during the study and nursing.
7. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
8. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only following a prophylactic regime.
9. Poorly controlled endocrine disorders, such as diabetes.
10. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
11. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
12. History of bleeding coagulopathies, or use of anticoagulants.
13. Use of isotretinoin (Accutane®) within six months prior to treatment or at physician discretion.
14. Treating over tattoo or permanent makeup.
15. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects undergoing breast reduction or breast mastectomy
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Independent blinded assessment | 6-months after treatment
  Independent blinded evaluator assessment of the surgical scar sites using the Global Aesthetic Improvement Scale (GAIS), comparing follow-up visit photographs for both the treated and untreated sides.
Principle Investigator (PI) evaluation of the scar(s) | 3- and 6-months after treatment
  PI evaluation of the scar(s) using the Manchester Scar Scale (MSS) at 3 and 6 months post-treatment for both the treated and untreated sides. Non-invasive skin assessments will be evaluated to document scar morphology, scar thickness/density and colorimetry for both the treated and untreated sides.

SECONDARY OUTCOMES:
Subject Satisfaction | 3- and 6-months after treatment
  Subject satisfaction of treatment using the Subject Satisfaction Scale
Histological Assessment | 1-, 3- and 6-months after treatment
  Histological assessment of the treated and the untreated (control) area.
Scar Morphology | Baseline, 3- and 6-months after treatment
  Scar morphology will be digitally analyzed using 3D photography camera
Ultrasonography | Baseline, 3- and 6-months after treatment
  High ultrasonography will be used to analyze scar thickness, epidermal thickness and skin density
Colorimetry | Baseline, 3- and 6-months after treatment
  o Colorimetry assessment will be used to establish a clinically acceptable objective assessment of patients' scars

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Department of Plastic Surgery, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan.